CLINICAL TRIAL: NCT02382458
Title: Developing the Dietary Inflammatory Index for Clinical Application
Acronym: IMAGINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Brie Turner-McGrievy, Associate Professor, University of South Carolina
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00037276
Record Dates: First submitted 2015-02-13; First posted 2015-03-06 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle intervention (Experimental): Participants will receive a year-long comprehensive, dietary, exercise, and stress management intervention. They will be asked to bring a partner of their choosing with them for support. The intervention will include a behavioral program to reduce inflammation.
  Interventions: Behavioral: Behavioral program to reduce inflammation
- Information intervention (Active Comparator): Participants will receive a year-long intervention that will involve receiving weekly (for the first 3 months) and then monthly (for the following 9 months) newsletters on cancer prevention and control (via e-mail or mail) that will provide the participant with information about cancer prevention and control strategies.
  Interventions: Behavioral: Newsletters on cancer prevention and control

INTERVENTIONS:
Behavioral: Newsletters on cancer prevention and control — E-mailed or mailed newsletters that provide information on how to prevent cancer
  Arms: Information intervention
Behavioral: Behavioral program to reduce inflammation — Group classes which will provide participants with information on achieving a healthy diet, increase physical activity, and manage stress
  Arms: Lifestyle intervention

SUMMARY:
Diet plays a central role in the regulation of chronic inflammation. However, until the investigators developed the dietary inflammatory index (DII) there had been no scientifically valid way to relate what individuals eat to the capacity of foods consumed to modulate inflammation. The DII provides a tool that will form the basis of a counseling/instructional system aimed at helping patients and their providers to control chronic, systemic inflammation by improving the diet with specific, actionable dietary recommendations, counseling, and expert instruction. The goal of this study is to test the applicability of a DII mobile tool and associated counseling measures in clinical practice.

DETAILED DESCRIPTION:
A large, persuasive, and ever-increasing body of evidence links chronic inflammation to virtually all of the chronic diseases that cause the majority of disability and death in the U.S., including diabetes, cardiovascular diseases (CVD), and cancer. Diet plays a central role in the regulation of chronic inflammation. However, until the investigators developed the dietary inflammatory index (DII) there had been no scientifically valid way to relate what individuals eat to the capacity of foods consumed to modulate inflammation. The new generation DII has now produced an impressive research base that ranges from predicting blood levels of inflammatory markers, to clinical conditions associated with inflammation, to a variety of health-related endpoints including cancer incidence, CVDs and mortality (several of which are already published). Connecting Health Innovations (CHI), LLC and the scientific and clinical research partners at the University of South Carolina are committed to translating these research findings to places of clinical need and public health relevance. That commitment to translation provides the motivation for the current proposal. The DII provides a tool that will form the basis of a counseling/instructional system aimed at helping patients and their providers to control chronic, systemic inflammation by improving the diet with specific, actionable dietary recommendations, counseling, and expert instruction. This project is part of Phase II of the grant, which includes: 1) Designing and implementing an intervention trial based on DII response associated recommendations aimed at reducing levels of chronic inflammation in two diverse populations in Columbia, South Carolina and 2) Providing data for developing methods for commercialization/ dissemination of the product and associated software.

ELIGIBILITY:
Inclusion Criteria:

* Are actively engaged as patients in the medical practices of University Specialty Clinics (under the direction of Dr. Victor Hirth) or Eau Claire Cooperative Health Care System (under the direction of Dr. Stuart Hamilton) or has physician consent
* Are ≥21 years of age;
* Are willing and able to participate fully in the study for a period of one year; and
* Are able to obtain travel to and from the intervention classes at the designated time.

Exclusion Criteria:

* Serious, unstable co-morbidity that would make participation in a diet and physical activity intervention difficult or risky including renal disease retinopathy, peripheral vascular disease or neuropathy;
* Any medications that are known to influence CRP levels such as chronic steroid (e.g., prednisone) use;
* Diagnoses of congestive heart failure, chronic renal failure, chronic liver disease (including alcoholic cirrhosis), cancer within the past year (except for non-melanoma skin cancer);
* Actively receiving cancer treatment;
* Have had any major surgeries in the past 3 months;
* Poor performance status according to the World Health Organization definitions (i.e., Level 3: symptomatic, >50% in bed, capable of only limited self-care; or Level 4: bedbound); or
* Life expectancy <3 years, on hospice, nursing home or other institutionalized care.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2015-05; Primary Completion 2017-02-28 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Markers of inflammation assessed via blood samples | 12 weeks
  C-reactive protein

SECONDARY OUTCOMES:
Changes in body weight assessed via digital scales | 52 weeks
Changes in dietary intake assessed via three 24-hour dietary recalls | 52 weeks
Markers of inflammation assessed via blood samples | 52 weeks
Changes in body composition assessed via DXA | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Brie Turner-McGrievy, Principal Investigator — University of South Carolina
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wirth MD, Turner-McGrievy G, Shivappa N, Murphy EA, Hebert JR. Interaction between Meal-timing and Dietary Inflammatory Potential: Association with Cardiometabolic Endpoints in a 3-month Prospective Analysis. J Nutr. 2023 Oct 28;153(12):3555-64. doi: 10.1016/j.tjnut.2023.10.023. Online ahead of print. PMID 39492485
- [Derived] Wirth MD, Jessup A, Turner-McGrievy G, Shivappa N, Hurley TG, Hebert JR. Changes in dietary inflammatory potential predict changes in sleep quality metrics, but not sleep duration. Sleep. 2020 Nov 12;43(11):zsaa093. doi: 10.1093/sleep/zsaa093. PMID 32406919
- [Derived] Turner-McGrievy GM, Wirth MD, Shivappa N, Dunn CG, Crimarco A, Hurley TG, West DS, Hussey JR, Hebert JR. Impact of a 12-month Inflammation Management Intervention on the Dietary Inflammatory Index, inflammation, and lipids. Clin Nutr ESPEN. 2019 Apr;30:42-51. doi: 10.1016/j.clnesp.2019.02.008. Epub 2019 Mar 1. PMID 30904228